CLINICAL TRIAL: NCT01752855
Title: A Phase 2b, Multicenter, Open-Label Study in Rheumatoid Arthritis Subjects Who Completed Preceding Study M13-390 With Adalimumab
Brief Title: Study in Rheumatoid Arthritis for Subjects Who Completed Preceding Study M13-390 With Adalimumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-692; 2012-003881-42 (EudraCT Number)
Record Dates: First submitted 2012-12-17; First posted 2012-12-19 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- New formulation of adalimumab 40 mg every other week (Experimental): New formulation adalimumab 40 mg every other week
  Interventions: Biological: New formulation adalimumab

INTERVENTIONS:
Biological: New formulation adalimumab — New formulation adalimumab 40 mg every other week
  Other Names: Humira

SUMMARY:
A Phase 2b, open-label extension (OLE) study in rheumatoid arthritis (RA) patients designed to collect long-term safety, tolerability, efficacy, and immunogenicity data of the proposed new adalimumab formulation.

DETAILED DESCRIPTION:
All participants who completed Study NCT01712178 had an opportunity to enroll into the study and to receive the new adalimumab formulation at a dose of 40 mg every other week (eow) for an additional 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has completed the preceding Study M13-390 for rheumatoid arthritis and has not developed any discontinuation criteria from that study.
2. If female, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy and/or hysterectomy) or is of childbearing potential and is practicing an approved method of birth control throughout the study and for 150 days after last dose of study drug. Examples of approved methods of birth control include the following (see local informed consent for more detail):

   * Condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD);
   * Hormonal contraceptives for 90 days prior to study drug administration;
   * A vasectomized partner.
3. Subjects must be able and willing to self-administer subcutaneous (SC) injections or have a qualified person available to administer SC injections.
4. Subject is judged to be in good general health as determined by the Principal Investigator based upon the results of medical history, physical examination, laboratory profile performed at Baseline.
5. Subjects must be able and willing to provide written informed consent and to comply with the requirements of this study protocol.

Exclusion Criteria:

1. Ongoing infections at Week 0 that have NOT been successfully treated. Subjects with ongoing infections undergoing treatment may be enrolled BUT NOT dosed until the infection has been successfully treated.
2. Subject currently uses or plans to use anti-retroviral therapy at any time during the study.
3. Subject plans to use any live vaccine during the study.
4. Positive pregnancy test at Baseline (Week 0).
5. Subject is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andy Payne, PhD, Study Director — AbbVie
Locations (20):
- United States (6):
  - Site Reference ID/Investigator# 92113, Mesa, Arizona
  - Site Reference ID/Investigator# 92118, Hemet, California
  - Site Reference ID/Investigator# 92117, Wichita, Kansas
  - Site Reference ID/Investigator# 92115, Clifton, New Jersey
  - Site Reference ID/Investigator# 92116, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 92114, Charleston, South Carolina
- Belgium (2):
  - Site Reference ID/Investigator# 92053, Brussels
  - Site Reference ID/Investigator# 92054, Liège
- Czechia (4):
  - Site Reference ID/Investigator# 91954, Brno
  - Site Reference ID/Investigator# 91955, Prague
  - Site Reference ID/Investigator# 91953, Uherské Hradiště
  - Site Reference ID/Investigator# 91956, Zlín
- Site Reference ID/Investigator# 92073, Ratingen, Germany
- Site Reference ID/Investigator# 92074, Vega Baja, Puerto Rico
- Romania (3):
  - Site Reference ID/Investigator# 92093, Bucharest
  - Site Reference ID/Investigator# 92095, Cluj-Napoca
  - Site Reference ID/Investigator# 92094, Ploieşti
- Slovakia (3):
  - Site Reference ID/Investigator# 92096, Banská Bystrica
  - Site Reference ID/Investigator# 92097, Senica
  - Site Reference ID/Investigator# 92098, Žilina

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA-approved. Please see US Prescribing Information for approved uses. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- New Formulation for 48 Weeks: New formulation of adalimumab 40 mg every other week for 24 weeks in Study NCT01712178, followed by 24 weeks of treatment with the new formulation of adalimumab 40 mg every other week
- Current Formulation for 24 Weeks, New Formulation for 24 Weeks: Current formulation of adalimumab 40 mg every other week for 24 weeks in Study NCT01712178, followed by 24 weeks of treatment with the new formulation of adalimumab 40 mg every other week
Period: Overall Study
Arm/Group | New Formulation for 48 Weeks | Current Formulation for 24 Weeks, New Formulation for 24 Weeks
Started | 44 | 44
Completed | 43 | 40
Not Completed | 1 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Withdrew Consent | 0 | 2
Not completed — Lack of Efficacy | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | New Formulation for 48 Weeks | Current Formulation for 24 Weeks, New Formulation for 24 Weeks | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (10.8) | 52.0 (12.0) | 53.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 74
  Male | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Disease Activity Score 28 (DAS28) at Weeks 36 and 48
Description: The Disease Activity Score (DAS28) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: Baseline (Study NCT01712178 Week 0 Visit), Weeks 36 and 48
Population: All available data were included. If a participant did not have a value for a given time of evaluation, but did have a value at times previous to this after the study drug treatment began, the last available value was used to replace the missing value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | New Formulation for 48 Weeks | Current Formulation for 24 Weeks, New Formulation for 24 Weeks
Number analyzed (Participants) | 44 | 44
units on a scale
  Week 36 | -2.4 (1.17) | -2.2 (1.05)
  Week 48 | -2.4 (1.29) | -2.2 (1.28)

2. Primary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 20 Response at Weeks 36 and 48
Description: American College of Rheumatology 20% (ACR20) response. A participant is a responder if the following 3 criteria for improvement from baseline are met:
  * ≥ 20% improvement in tender joint count;
  * ≥ 20% improvement in swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters:
    * Physician global assessment of disease activity
    * Patient global assessment of disease activity
    * Patient assessment of pain
    * Disability Index of the Health Assessment
    * CRP (Acute phase reactant (Erythrocyte sedimentation rate/C-reactive protein))
Time Frame: Baseline (Study NCT01712178 Week 0 Visit), Weeks 36 and 48
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | New Formulation for 48 Weeks | Current Formulation for 24 Weeks, New Formulation for 24 Weeks
Number analyzed (Participants) | 44 | 44
percentage of participants
  Week 36 | 72.7 | 76.7
  Week 48 | 74.4 | 80.0

3. Primary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 50 Response at Weeks 36 and 48
Description: American College of Rheumatology 50% (ACR50) response. A participant is a responder if the following 3 criteria for improvement from baseline are met:
  * ≥ 50% improvement in tender joint count;
  * ≥ 50% improvement in swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
    * Physician global assessment of disease activity
    * Patient global assessment of disease activity
    * Patient assessment of pain
    * Disability Index of the Health Assessment
    * CRP (Acute phase reactant (Erythrocyte sedimentation rate/C-reactive protein))
Time Frame: Baseline (Study NCT01712178 Week 0 Visit), Weeks 36 and 48
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | New Formulation for 48 Weeks | Current Formulation for 24 Weeks, New Formulation for 24 Weeks
Number analyzed (Participants) | 44 | 44
percentage of participants
  Week 36 | 50.0 | 51.2
  Week 48 | 53.5 | 57.5

4. Primary Outcome: Mean Change From Baseline in Health Assessment Questionnaire (HAQ-DI) at Weeks 36 and 48
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. The minimal clinically important difference (MCID) defined for the HAQ-DI is 0.22. HAQ remission indicating normal physical function is defined by HAQ-DI < 0.5.
Time Frame: Baseline (Study NCT01712178 Week 0 Visit), Weeks 36 and 48
Population: Data from participants receiving the new formulation of adalimumab in Study NCT01712178 were analyzed for 44 and 43 participants, respectively, at weeks 36 and 48. Data for the participants receiving the current formulation of adalimumab in Study NCT01712178 were analyzed for 43 participants at week 36 and 40 participants at week 48.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | New Formulation for 48 Weeks | Current Formulation for 24 Weeks, New Formulation for 24 Weeks
Number analyzed (Participants) | 44 | 43
units on a scale
  Week 36 | -0.5 (0.60) | -0.5 (0.69)
  Week 48 | -0.5 (0.57) | -0.5 (0.58)

5. Secondary Outcome: Percentage of Participants Positive for Anti-adalimumab Antibody
Description: Percentage of participants with anti-adalimumab antibody
Time Frame: Week 24 through Week 48
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | New Formulation for 48 Weeks | Current Formulation for 24 Weeks, New Formulation for 24 Weeks
Number analyzed (Participants) | 44 | 44
percentage of participants | 13.6 | 18.2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of study drug administration until 70 days following the last dose, approximately 58 weeks. Serious adverse events were collected from the time the participant signed the informed consent.
Arm/Group | New Formulation for 48 Weeks | Current Formulation for 24 Weeks, New Formulation for 24 Weeks
Serious Adverse Events (participants affected / at risk) | 2/44 | 1/44
Other Adverse Events (participants affected / at risk) | 18/44 | 19/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | New Formulation for 48 Weeks (N=44) | Current Formulation for 24 Weeks, New Formulation for 24 Weeks (N=44)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | New Formulation for 48 Weeks (N=44) | Current Formulation for 24 Weeks, New Formulation for 24 Weeks (N=44)
DYSPEPSIA (Gastrointestinal disorders) | 3 | 3
CYSTITIS (Infections and infestations) | 4 | 2
NASOPHARYNGITIS (Infections and infestations) | 6 | 7
ORAL HERPES (Infections and infestations) | 3 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 4
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 3
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 | 4
HEADACHE (Nervous system disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.